CLINICAL TRIAL: NCT05437094
Title: A Phase 1, Open-Label, Fixed Sequence Study to Investigate the Effect of Coadministration of Itraconazole on the Pharmacokinetics of CRD-740 in Healthy Adult Subjects
Brief Title: Effect of Coadministration of Itraconazole on the Pharmacokinetics of CRD-740
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Cardurion Pharmaceuticals, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: CRD-740-101
Record Dates: First submitted 2022-06-17; First posted 2022-06-29 (Actual); Last update posted 2025-05-15 (Actual); Status verified 2023-02

CONDITIONS: Clinical Pharmacology; Pharmacokinetics; Cardiovascular Diseases; Heart Failure
MeSH Terms: conditions — Cardiovascular Diseases; Heart Failure | interventions — Itraconazole

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- CRD-740 (Other): CRD-740 single dose administered alone
  Interventions: Drug: CRD-740
- CRD-740 and Itraconazole (Other): CRD-740 single dose administered with Itraconazole
  Interventions: Drug: CRD-740; Drug: Itraconazole

INTERVENTIONS:
Drug: CRD-740 — CRD-740
Drug: Itraconazole — Itraconazole
  Arms: CRD-740 and Itraconazole

SUMMARY:
This is a Phase 1, single-site, open-label, fixed sequence crossover study to investigate the effect of coadministration of itraconazole on the pharmacokinetics of CRD-740 in healthy male and female subjects. Subjects will be admitted into the study site on Day -1 and will be confined to the study site until discharge on Day 16. Subjects will receive CRD-740 orally on Days 1 and 10. Itraconazole will be given once daily, orally, on Days 7 through 15.

ELIGIBILITY:
Inclusion Criteria:

1. Males or females, of any race, between 18 and 55 years of age, inclusive.
2. Body mass index between 18.0 and 32.0 kg/m2, inclusive.
3. In good health, determined by no clinically significant findings as assessed by the investigator.
4. Adhere to all contraception criteria.

Exclusion Criteria:

1. Significant medical history as determined by the investigator.
2. History of significant hypersensitivity, intolerance, or allergy to any drug compound, food, or other substance, including itraconazole, unless approved by the investigator (or designee).
3. History of stomach or intestinal surgery or resection that would potentially alter absorption or excretion of orally administered drugs (uncomplicated appendectomy and hernia repair will be allowed).
4. Any clinically significant abnormalities in clinical chemistry, hematology, or urinalysis results, as judged by the investigator.
5. History or presence of an abnormal ECG.
6. Use or intend to use any medications/products/herbal remedies known to alter drug absorption, metabolism, or elimination processes, including St. John's wort, within 30 days prior to check-in, unless deemed acceptable by the investigator (or designee).
7. Drugs affecting CYP3A4 should be refrained from use for 3 weeks, or 5 half-lives (whichever is longer), prior to check-in through to follow-up.
8. Positive urine drug screen at screening or positive alcohol breath test result or positive urine drug screen at check-in.21. History of alcoholism or drug/chemical abuse within 12 months prior to check-in.
9. Ingestion of poppy seed, Seville orange, or grapefruit containing foods or beverages within 7 days prior to check-in.

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 20 (Actual)
Dates: Start 2022-06-27 (Actual); Primary Completion 2022-08-03 (Actual); Study Completion 2022-08-10 (Actual)

PRIMARY OUTCOMES:
AUC0-24 of CRD-740 alone and with coadministration of itraconazole | Day 1 to Day 16
AUC0-inf of CRD-740 alone and with coadministration of itraconazole | Day 1 to Day 16
AUC0-t of CRD-740 alone and with coadministration of itraconazole | Day 1 to Day 16
Cmax of CRD-740 alone and with coadministration of itraconazole | Day 1 to Day 16

SECONDARY OUTCOMES:
Half life (t1/2) of CRD-740 | Day 1 to Day 16
Time to maximum concentration (Tmax) of CRD-740 | Day 1 to Day 16
Oral clearance (CL/F) of CRD-740 | Day 1 to Day 16
Apparent volume of distribution during terminal phase (Vz/F) of CRD-740 | Day 1 to Day 16

CONTACTS AND LOCATIONS:
Locations (1):
- Cardurion Investigative Site, Dallas, Texas, United States

IPD SHARING:
Plan to Share IPD: No